CLINICAL TRIAL: NCT06817668
Title: Evaluating Tolerability of Elective Pelvic Ultra Hypofractionated Irradiation Treatment (ePUHRT) With High Dose Rate Brachytherapy Boost for Unfavorable and Higher Risk Prostate Cancer
Brief Title: Evaluating Tolerability of ePUHRT With Brachytherapy Boost
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Omar Ishaq, Assistant Professor of Clinical Urology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0832
Record Dates: First submitted 2024-10-09; First posted 2025-02-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Brachytherapy boost
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ePURT 5Gy x 5 fractions with single HDR boost of 15Gy (Experimental): Single arm non-randomized non-inferiority study exploring tolerability of ePURT 5Gy x 5 fractions delivered on noncontiguous weekdays with single HDR boost of 15Gy.
  Interventions: Radiation: ePURT 5Gy x 5 fractions with single HDR boost of 15Gy

INTERVENTIONS:
Radiation: ePURT 5Gy x 5 fractions with single HDR boost of 15Gy — ePURT 5Gy x 5 fractions delivered on noncontiguous weekdays with single HDR boost of 15Gy.

SUMMARY:
The purpose of this study is to evaluate the tolerability and toxicity of combining two radiation therapy methods for prostate cancer: Elective Pelvic Ultra Hypofractionated Irradiation Treatment (ePUHRT), which is an external beam radiotherapy with High Dose Rate Brachytherapy Boost (form of internal radiation where a cancer doctor implants a small plastic tube or balloon (catheter) in the tumor).

DETAILED DESCRIPTION:
Progression free survival from irradiation dose escalation has been demonstrated across multiple prospective randomized studies. Irradiation dose escalation delivered by dual therapy (consisting of external beam irradiation treatment with brachytherapy boost, a type of internal radiation) offers improved survival. Brachytherapy boost makes it possible to safely deliver higher irradiation dose to the prostate gland than can be achieved with dose escalation by standard fractionated external beam treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Capable of providing informed consent and HIPAA authorization
3. Karnofsky performance score ≥ 70
4. Pathologically confirmed unfavorable intermediate, high, and very high-risk prostate cancer per treating physician
5. Candidate plans to undergo the standard of care prostate high dose brachytherapy boost procedure

Exclusion Criteria:

1. Prior pelvic irradiation treatment
2. Prior rectal surgery which precludes instrumentation with rectal ultrasound probe.
3. Evidence of nodal or distant disease on screening diagnostic work up.
4. Prior prostatectomy, Holmium laser enucleation of the prostate or transurethral resection of the prostate procedure
5. International Prostate Symptom Score (IPSS) score > 16 despite medical therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with acute grade ≥ 2 GU toxicity | 3 months
  Physician-reported acute grade ≥ 2 GU toxicity at 3 months post ePUHRT with HDR boost measured by CTCAE version 5.

SECONDARY OUTCOMES:
Percentage of participants with acute grade ≥ 2 GI toxicity | 3 months
  Acute grade ≥ 2 GI toxicity at 3 months post ePUHRT with HDR boost by CTCAE version 5
Percentage of participants with acute grade ≥ 2 GU toxicity | 3 months
  Self-reported acute grade ≥ 2 GU toxicity at 3 months post ePUHRT with HDR boost measured by PRO-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ishaq, MD, Principal Investigator — Indiana University Simon Comprehensive Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided